CLINICAL TRIAL: NCT01171781
Title: A Randomized Phase II Study of Concurrent Chemoradiation With Every 3 Week of Cisplatin vs With Weekly Cisplatin in Locally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myung-Ju Ahn, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-09-037
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Nasophayngeal Carcinoma Between Stage II and IVb
MeSH Terms: interventions — Cisplatin

ARMS (2):
- 3 weekly CDDP based CCRT (Active Comparator): radiation (conventioal or IMRT) with 3 cycles of 3-weekly cisplatin
  Interventions: Drug: cisplatin (3 weekly)
- weekly cisplatin based CCRT (Experimental): radiation (conventional or IMRT) with 7 cycles of weekly cisplatin therapy
  Interventions: Drug: cisplatin (weekly)

INTERVENTIONS:
Drug: cisplatin (3 weekly) — radiation with cisplatin (100mg/m2) on D1,D22,D43 and followed by adjuvant chemotherapy (3 cycles of FP)
  Arms: 3 weekly CDDP based CCRT
Drug: cisplatin (weekly) — radiation with 7 cycles of cisplatin (40mg/m2) on D1,8,15,22,29,36,43, and followed by adjuvant chemothrapy (FP X3)
  Arms: weekly cisplatin based CCRT

SUMMARY:
The study try to show the weekly cisplatin based CCRT is not inferior to 3-weekly cisplabe based CCRT in terms of 3-yr progression free survival rate in advanced nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed nasopharyngeal carcinoma age of 18 years or over stage II ~ IVb no history of chemotherapy, radiotherapy, or immunotherapy for NPC with measurable lesion based on RECIST 1.1 ECOG PS 0 ~2 good organ function (liver, renal, hematologic)

Exclusion Criteria:

* active infectious disease requiring antibiotics uncontrolled heart disease pregnancy and on feeding state history of other malignancy within 5 years before enrollment, except for well treated non-melanomatous skin cancer, in situ cervical cancer, thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival rate at 3 years | 36 months

SECONDARY OUTCOMES:
overall survival rate | 36 months
objective response rate | 36 months
toxicity | 36 months
quality of life | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea